CLINICAL TRIAL: NCT01146639
Title: Usefulness of DynaCT Compared to Multidetector CT as Preoperative Imaging Before Insertion of Aortic Stentgraft.
Brief Title: DynaCT in Preoperative Imaging Before Insertion of Stentgraft
Acronym: DynaCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: rek 4.2008.802
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: EVAR DynaCT
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — iodixanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MDCT and additional DynaCT (Experimental)
  Interventions: Radiation: DynaCT; Drug: Iodixanol

INTERVENTIONS:
Radiation: DynaCT — One extra set of images with DynaCT including one extra injection of contrast medium.
Drug: Iodixanol — One extra set of images with DynaCT including one extra injection of 50 ml contrast medium.
  Other Names: Visipaque Amersham Health 270 mg I/ml

SUMMARY:
Endovascular therapy of Aortic Aneurysms depends on good imaging facilities. A relatively new kind of x-ray equipment makes it possible to create computer tomography (CT) - like slice images in the operating room. The purpose of this study is to verify the clinical usefulness of DynaCT in a preoperative setting. To do so we compare aortic measurements in DynaCT to the same measurements in ordinary CT-images which are regarded the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Not inserted stent graft before.
* Patiens over 60 Years old.
* Able to give informed consent.

Exclusion Criteria: Not

-

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-08; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Verify clinical usefulness of DynaCT images in preoperative imaging. | One year

CONTACTS AND LOCATIONS:
Locations (1):
- St Olavs Hospital, Operating Room of the Future., Trondheim, Norway

REFERENCES:
- [Result] Eide KR, Odegard A, Myhre HO, Hatlinghus S, Haraldseth O. DynaCT in pre-treatment evaluation of aortic aneurysm before EVAR. Eur J Vasc Endovasc Surg. 2011 Sep;42(3):332-9. doi: 10.1016/j.ejvs.2011.05.014. Epub 2011 Jul 22. PMID 21782483